CLINICAL TRIAL: NCT00374114
Title: A Pilot Study to Evaluate Ultrasonic Surgical Aspiration as a Treatment Modality for Cervical Dysplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Integra LifeSciences Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: d34c09
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2008-12-15 (Estimated); Status verified 2008-12

CONDITIONS: Cervical Dysplasia
Keywords: cervical; dysplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Conization

INTERVENTIONS:
Procedure: cervical conization
Procedure: ultrasonic surgical aspiration of the cervix

SUMMARY:
Ultrasonic surgical aspiration of the cervix may be an effective method of treating cervical dysplasia without compromising the integrity of the cervix in reproductive age women.

DETAILED DESCRIPTION:
Women age 18 to 55 years of age with Cervical Intraepithelial Neoplasia 2 or 3 on colposcopy with a negative EndoCervical Curettage are enrolled in a pilot study comparing ultrasonic surgical aspiration and traditional cervical excision procedure for the treatment of cervical dysplasia. In this pilot study, the patients serve as their own control group. Prior to receiving the traditional treatment for cervical dysplasia consisting of Cold Knife Conization with EndoCervical Curettage, each patient's cervix is treated with ultrasonic surgical aspiration. The aspirate is sent to pathology and the results compared with the findings from the cervical cone biopsy. The patients then are followed with Liquid-based Cytology pap smears every 4 to 6 months until completion of the study enrollment/treatment period.

ELIGIBILITY:
Inclusion Criteria:

* cervical intraepithelial neoplasia II or III
* negative endocervical curettage
* not pregnant
* cervical conization is part of treatment plan

Exclusion Criteria:

* positive endocervical curettage
* pregnant
* medically unable to undergo surgery

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Adequate treatment of cervical dysplasia

CONTACTS AND LOCATIONS:
Overall Officials: Stephen DePasquale, DO, Principal Investigator — University of Tennessee
Locations (2):
- United States (2):
  - University of Tennessee College of Medicine, Chattanooga, Tennessee
  - University of Tennessee Health Sciences Center, Memphis, Tennessee